CLINICAL TRIAL: NCT00912886
Title: Neuroactive Steroids and Cognition in Humans: Pregnenolone Sulfate an Early Marker of the Memory Loss Associated With Alzheimer's Disease
Brief Title: Pregnenolone Sulfate an Early Marker of the Memory Loss in Alzheimer's Disease
Acronym: STERMEM
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: P071237
Record Dates: First submitted 2009-06-02; First posted 2009-06-03 (Estimated); Last update posted 2013-04-11 (Estimated); Status verified 2013-04

CONDITIONS: Alzheimer Disease
Keywords: alzheimer; memory; neurosteroids
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma and serum from AD patients and from Controls
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Case: Patients with early and moderate AD
- 2: Controls: AD free volunteer-controls matched for gender and age

SUMMARY:
The steroid pregnenolone sulfate (PREGS) may be one of the factors responsible for the memory decline related to normal aging or associated with Alzheimer's disease (AD). The purpose of this study is to determine whether plasma levels of PREGS are decreased patients with at mild to moderate AD compared with AD-free control subjects matched for gender and age and to see whether they are inversely correlated with the severity of memory deficits in AD patients. The hypothesis is that blood levels of PREGS are decreased with advanced age and with the stage of AD that would be positively correlated with memory deficits. Therefore PREGS could be considered as an early marker of the memory deficits in AD.

DETAILED DESCRIPTION:
PREGS is a derivative of pregnenolone which the obligatory precursor of all steroid hormones originating from the gonads and adrenal glands. In rodents, PREGS has been demonstrated to improve memory performance in various behavioural tests. In humans, PREGS is one the most abundant circulating steroids. There are some indications about its decrease in blood during aging, and in brain samples from aged patients with AD, low concentrations of PREGS have been correlated with high levels of beta-amyloid peptide and phosphorylated tau protein. To date, a precise and rigorous evaluation of PREGS blood concentrations during aging is lacking and the relationship between these concentrations and the memory loss associated with AD has not been established.

Primary objective To show that plasma concentrations of PREGS are decreased in AD patients (" case ") compared to free-AD subjects (" controls "), matched for gender and age.

Secondary objectives

* To show that plasma concentrations of PREGS are inversely correlated with the severity of memory deficits in AD patients.
* To show that plasma concentrations of PREGS are correlated with the memory scores in the controls.
* To show that plasma concentrations of PREGS decrease in the controls.
* To search for a relationship between some of PREGS metabolites and age or the severity of memory deficits.

This is a case-control study that will comprise 200 subjects aged over 70 years, including 100 outpatients with mild to moderate AD and 100 AD-free volunteer controls matched on age and gender. These two groups will be stratified into age-sub-groups [70-74] [75-79] [80-84] [85-89] > 90 years and will include 10 men and 10 women per sub-group.

AD patients and controls will be enrolled and evaluated in the geriatric centres of 5 hospitals namely BICETRE, BROCA, PAUL BROUSSE, PITIE-SALPETRIERE and ROTHSCHILD. They will all be submitted to a clinical examination, biological analyses, cognitive tests and a brain magnetic resonance imaging scan. Blood will be collected from all subjects for steroid analysis by gas chromatography-mass spectrometry, a sensitive and accurate methodology that allows simultaneous quantification of several steroids in the same individual sample. PREGS and some of its metabolites will be identified and quantified at the "Institute medical of heath" (INSERM U788).

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged over 70 years who have signed informed consent for participation to the study and are affiliated to a social security regimen.
* For patients: subjects with probable AD according to the DSM-IV criteria and the NINCDS/ADRDA criteria and with mild to moderate probable AD: MMSE score> 15.
* For Controls: subjects without cognitive deficits on neuropsychological tests: scores of MMSE > 26 and of the 5 Word test equal to 10/10 and of the Clock Drawing test equal to 7/7.

Exclusion Criteria:

* Guardianship
* History of cerebrovascular disease, Parkinson's disease, other known dementia, epilepsy
* Major depression
* Serious sensory disorders; deficits in language & comprehension
* Serious heart or hepatic insufficiencies, renal or respiratory failures
* Unstable diabetes or endocrine disorders, thyroid dysfunction, cancer, inflammatory syndrome, malnutrition
* Cognitive training during the 6 previous months
* Medications: steroids (HRT, androgens, corticoids), anti-depressants, cholinesterase inhibitors, thyroid hormones, synthetic anti-thyroids
* Contraindications for MRI: metallic implants & claustrophobia

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: * AD Patients will be recruited among the new patients from the consultations of the geriatric centres involved in the study
  * Controls will be recruited from the consultations, associations of aged persons or among the relatives of the patient
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2009-09; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Plasma concentrations of PREGS determined by GC-MS | At the day of diagnostic blood collection

SECONDARY OUTCOMES:
Memory scores of the RL-RI test according to the GROBER and BUSCKE test | At the day of blood collection
Plasma concentrations of PREGS metabolites | At the day of blood collection

CONTACTS AND LOCATIONS:
Overall Officials: Sebastien Weill-Engerer, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris Hôpital Rothschild; Yvette Akwa, PhD, Study Director — INSERM U788
Locations (6):
- France (6):
  - Assistance publique - Hôpitaux de Paris Hôpital Bicêtre, Le Kremlin-Bicêtre
  - Inserm Umr 788, Le Kremlin-Bicêtre
  - AP-HP Hôpital Rothschild, Paris
  - Assistance Publique - Hôpitaux de Paris Hôpital Broca, Paris
  - Assistance Publique - Hôpitaux de Paris, Hôpital Pitié-Salpétrière, Paris
  - Assistance Publique - Hôpitaux de Paris, Hôpital Paul Brousse, Villejuif